CLINICAL TRIAL: NCT02374866
Title: Monitoring Obese Patients: Impact on the Frequency of Monitoring Weight, Quality of Life, Dietary Behavior, Physical Ability and Comorbidities
Brief Title: Monitoring Obese Patients : Impact on the Frequency of Monitoring Weight
Acronym: SUIVIOBESITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I13031 SUIVI OBESITE
Record Dates: First submitted 2015-02-18; First posted 2015-03-02 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; Morbid Obesity; Quality of Life
Keywords: Obesity; Morbid Obesity; Therapeutic education
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional monitoring (No Intervention): The control group will follow the current center: every four months for a year, combined with monitoring by email or regular mail during the year.
- Closer monitoring (Experimental): The experimental group will follow a closer monitoring than the control group : every two months for one year in,stead of every 4 months for a year.
  Follow by email or mail is identical to the control group.
  Interventions: Other: closer monitoring

INTERVENTIONS:
Other: closer monitoring
  Arms: Closer monitoring

SUMMARY:
The literature data show that long-term monitoring has an effect on weight loss, comorbidity and on improving the quality of life. However, there are still no studies on monitoring obese patients after taking initial multidisciplinary approach. The recommendations of the HAS 2011 advocated "continuous monitoring needed to prevent weight regain, monitor the consequences of overweight and treat comorbidities. This requires a long-term support. "The frequency of follow-up consultations is not specified and "must be adapted to achieve a weight loss target and maintain." Having no specific recommendations on the frequency of monitoring, the investigators chose to experiment closer monitoring than our current monitoring to assess what is the best frequency monitoring, in terms of: weight loss, quality of life, feeding behavior, changes in physical abilities, evolution of comorbidities associated with obesity. The recommendations of the HAS 2011 advocate support of a multidisciplinary obesity for weight loss of 5% to 10 %, which, if maintained, can reduce comorbidities associated with obesity (type 2 diabetes, hypertension, pain associated with osteoarthritis).

DETAILED DESCRIPTION:
2 groups of randomized patients will be followed:

* The control group will follow the current center: every four months for a year, combined with monitoring by email or regular mail during the year.
* The experimental group will be a follow-up every two months for one year HDJ more of the same followed by email or postal mail.

Follow by email or mail is identical to the control group, as well as HDJ 12 months.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 - ≤ 75 years
* Obesity with a BMI ≥ 35 or ≥ 30 if associated with at least one comorbidity whose support was commenced or continued during the initial hospitalization.
* Patients hospitalized for a period of at least 3 weeks in the Bernard Descottes center and were supported on dietary, psychological, psychomotor and physical education in a therapeutic approach.
* Patients who have signed consent form.
* Patients who never underwent bariatric surgery and bariatric surgery have not seen in the year following their hospitalization in Bernard Descottes Center.
* Patient accepting the constraints of the protocol in case of close monitoring.
* Patients able to travel with their own vehicle to Bernard Descottes Center.
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* - Patients who have hospitalized in Bernard Descottes Center.
* Failure to follow the protocol because of insufficient command of French or concomitant illness.
* Pregnant or breastfeeding.
* Patients under guardianship or under judicial protection.
* Participation to another trial which can impact on patient's experimental disease during all the study, and patients who are in an exclusion period of another trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
percentage of weight loss at 12 months | 1 year
percentage of change in BMI at 12 months | 1 year

SECONDARY OUTCOMES:
Change of waist at 12 months | 1 year
Changes in body composition | 1 year
Change of quality of life at 12 months | 1 year
Change of medication at 12 months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cécile de Rouvray, Md, Principal Investigator — Centre de l'Obesite Bernard Descottes
Locations (1):
- Centre de suivi de l'obésite Bernard Descottes, Saint-Yrieix-la-Perche, France